CLINICAL TRIAL: NCT06957353
Title: Oblique Sliding K-wire Technique For Controlling Calcaneal Displacement Osteotomy In Flat Foot Correction
Brief Title: Oblique K-wire Control in Calcaneal Osteotomy for Flatfoot Correction
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mina S. Fekry, assistant lecturer, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AUH-Calcaneal_osteotomy-2025
Record Dates: First submitted 2025-04-21; First posted 2025-05-04 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Flat Foot
Keywords: flat foot; calcaneal osteotomy
MeSH Terms: conditions — Flatfoot

STUDY DESIGN:
Intervention Model Description: using an oblique K-wire technique in controlling Calcaneal displacement during osteotomy in flatfoot correction
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Oblique K-wire Control in Calcaneal Osteotomy for Flatfoot Correction (Other): oblique K-wire technique in controlling Calcaneal displacement during osteotomy in flatfoot correction
  Interventions: Procedure: oblique K-wire technique in controlling Calcaneal displacement during osteotomy in flatfoot correction

INTERVENTIONS:
Procedure: oblique K-wire technique in controlling Calcaneal displacement during osteotomy in flatfoot correction — Under spinal Anaesthesia , patients will placed in lateral decubitus position. A standard lateral incision will be made over the calcaneus, and the osteotomy site will be exposed. An oblique K-wire will be inserted percutaneously into the posterior calcaneus under fluoroscopic guidance to facilitate the desired displacement. Cannulated screws will then be inserted across the osteotomy site to secure the calcaneal fragment. Post-operative care will include a non-weight bearing protocol for six weeks, followed by gradual weight bearing as tolerated.

SUMMARY:
Adult-acquired flatfoot deformity (AAFD) often requires surgical correction when conservative methods fail. Calcaneal displacement osteotomy is a key procedure in restoring alignment. This study introduces a novel K-wire technique to enhance control during surgery and minimize complications related to manual manipulation. It builds on prior research highlighting the limitations of traditional approaches in achieving precise fragment positioning.

DETAILED DESCRIPTION:
Flat foot deformity, particularly adult - acquired flatfoot (AAFD), often necessitates surgical intervention when conservative treatment fail. Calcaneal displacement osteotomy is a common surgical procedure for correcting calcaneal displacement and achieving stable fixation. The proposed K-wire technique offers a novel approach to improve control and reduce complications associated with manual manipulation during surgery. Previous studies have indicated challenges with traditional methods in achieving precise fragment control. This study aims to address these gaps.

ELIGIBILITY:
Inclusion Criteria:

* symptomatic flatfoot that will undergo flatfoot correction with calcaneal displacement osteotomy.

Exclusion Criteria:

* prior foot surgery
* Severe comorbidities or contradictions of the surgery

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
assessment of degree of desired displacement | baseline
  Intra-operative assessment of degree of desired displacement clinical and radiological

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Mostafa Kotb, professir, Principal Investigator — Assiut University
Locations (1):
- Assiut University Hospital, Asyut, Egypt

REFERENCES:
- [Background] Cai Y, Zhao Z, Huang J, Yu Z, Jiang M, Kang S, Yuan X, Liu Y, Wu X, Ouyang J, Li W, Qian L. Morphological changes in flatfoot: a 3D analysis using weight-bearing CT scans. BMC Med Imaging. 2024 Aug 19;24(1):219. doi: 10.1186/s12880-024-01396-0. PMID 39160476
- [Background] Brilhault J. Calcaneal osteotomy for hindfoot deformity. Orthop Traumatol Surg Res. 2022 Feb;108(1S):103121. doi: 10.1016/j.otsr.2021.103121. Epub 2021 Oct 20. PMID 34687951
- [Background] Mueller G, Frosch KH, Barg A, Schlickewei C, Weel H, Krahenbuhl N, Priemel M, Mueller E. Impact of the medial displacement calcaneal osteotomy on foot biomechanics: a systematic literature review. Arch Orthop Trauma Surg. 2024 May;144(5):1955-1967. doi: 10.1007/s00402-024-05267-9. Epub 2024 Mar 30. PMID 38554203